CLINICAL TRIAL: NCT03257852
Title: A Phase 2a, Randomized, Placebo-Controlled, Double-Blind, Parallel Group Study to Evaluate the Efficacy and Safety of ASP5094 in Patients With Rheumatoid Arthritis on Methotrexate
Brief Title: A Study to Evaluate the Efficacy and Safety of ASP5094 in Patients With Rheumatoid Arthritis on Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5094-CL-0201
Record Dates: First submitted 2017-08-20; First posted 2017-08-22 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Methotrexate; Arthritis, Rheumatoid; ASP5094
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASP5094 Group (Experimental): To be intravenously administered ASP5094 in patients with rheumatoid arthritis (RA) treated with methotrexate.
  Interventions: Drug: ASP5094; Other: Methotrexate therapy
- Placebo Group (Placebo Comparator): To be intravenously administered ASP5094 in patients with rheumatoid arthritis (RA) treated with methotrexate.
  Interventions: Drug: Placebo; Other: Methotrexate therapy

INTERVENTIONS:
Drug: ASP5094 — intravenously administration
  Arms: ASP5094 Group
Drug: Placebo — intravenously administration
  Arms: Placebo Group
Other: Methotrexate therapy — MTX must have been continuously orally administered for at least 90 days prior to screening, with stable dosage for at least 28 days prior to screening, and will be continuously administered with the same dosage throughout the study period.

SUMMARY:
The objective of this study is to evaluate the efficacy, safety and pharmacokinetics of ASP5094 in patients with rheumatoid arthritis (RA) treated with background methotrexate (MTX).

DETAILED DESCRIPTION:
The study drug will be intravenously administered.

ELIGIBILITY:
Inclusion Criteria:

* Subject has RA diagnosed according to the 1987 American College of Rheumatology (ACR) criteria or the 2010 ACR/European League Against Rheumatism (EULAR) criteria at least 6 months prior to screening.
* Subject meets the 1991 ACR Revised Criteria for the Classification of Global Functional Status in RA Class I, II, or III at screening.
* At screening and baseline, subject has active RA as evidenced by both of the following:

  * ≥ 6 tender/painful joints (using 68-joint assessment)
  * ≥ 6 swollen joints (using 66-joint assessment)
* Subject meets the criterion for a CRP level (Latex Agglutination method) at screening.
* Subject who has continuously received Methotrexate for at least 90 days prior to screening and who is able to continue a stable dose of Methotrexate from at least 28 days prior to screening throughout the study period.

Exclusion Criteria:

* Subject has deviated from the criteria for previous and concomitant treatment before baseline.
* Subject has an ongoing infection requiring antibiotics.
* Subject is determined to be an inadequate responder to a prior biologic disease modifying antirheumatic drugs (DMARDs) or Janus kinase (JAK) inhibitors.
* Subject has participated in previous ASP5094 clinical trial.
* Subject has participated in a clinical trial or post-marketing clinical study of another ethical drug or medical device within 12 weeks (84 days).
* Subject has another inflammatory arthritis than RA, or any other articular symptom which may affect on joint assessment.
* Subject meets any of the criteria for laboratory values at screening.
* Subject has a positive T-SPOT or QuantiFERON Gold test within 90 days prior to screening or at screening.
* Subject has a history of or concurrent malignant tumor.
* Subject has autoimmune disease except for RA or any severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, neurological, or mental illness.
* Subject has a history of clinically significant allergy.
* Subject has clinically significant abnormalities on 12-lead electrocardiogram (ECG) at screening.
* Subject has a history of Human Immunodeficiency Virus (HIV) infection.
* Subject had surgery within 30 days prior to screening or has a planned elective surgery.
* Subject has a wound that is currently healing at baseline.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
ACR50 response rate | Week 12
  To assess ACR (American College of Rheumatology) 50 for efficacy

SECONDARY OUTCOMES:
ACR50 response rate | Up to Week 16
  To assess ACR (American College of Rheumatology) 50 for efficacy
ACR20 response rate | Up to Week 16
  To assess ACR (American College of Rheumatology) 20 for efficacy
ACR70 response rate | Up to Week 16
  To assess ACR (American College of Rheumatology) 70 for efficacy
Change from baseline in DAS28-CRP score | Baseline and Up to Week 16
  To assess DAS28-CRP (Disease Activity Score28 - C-reactive protein) for efficacy
Change from baseline in DAS28-ESR score | Baseline and Up to Week 16
  To assess DAS28-ESR (Disease Activity Score28 - Erythrocyte sedimentation rate) for efficacy
Change from baseline in Tender Joint Count (68 joints) | Baseline and Up to Week 16
  To assess Tender Joint Count for efficacy
Change from baseline in Swollen Joint Count (66 joints) | Baseline and Up to Week 16
  To assess Swollen Joint Count for efficacy
Percentage of subjects achieving DAS28-CRP score for remission (<2.6) | Up to Week 16
  To assess DAS28-CRP score for efficacy
Percentage of subjects achieving DAS28-ESR score for remission (<2.6) | Up to Week 16
  To assess DAS28-ESR score for efficacy
Percentage of subjects achieving DAS28-CRP score for low disease activity (≦3.2) | Up to Week 16
  To assess DAS28-CRP score for efficacy
Percentage of subjects achieving DAS28-ESR score for low disease activity (≦3.2) | Up to Week 16
  To assess DAS28-ESR score for efficacy
Change from baseline in CRP | Baseline and Up to Week 16
  To assess CRP (C-reactive protein) for efficacy
Change from baseline in ESR | Baseline and Up to Week 16
  To assess ESR (Erythrocyte sedimentation rate) for efficacy
Percentage of subjects achieving EULAR response criteria of "Good Response" | Up to Week 16
  To assess EULAR (European league Against Rheumatism) response criteria for efficacy
Percentage of subjects achieving EULAR response criteria of "Good Response" or "Moderate Response" | Up to Week 16
  To assess EULAR response criteria for efficacy
Percentage of subjects achieving ACR/EULAR score for remission | Up to Week 16
  To assess ACR/EULAR remission for efficacy
Percentage of subjects achieving SDAI score ≦ 3.3 (SDAI remission) | Up to Week 16
  To assess SDAI (Simplified Disease Activity Index) score for efficacy
Percentage of subjects achieving CDAI score ≦ 2.8 (CDAI remission) | Up to Week 16
  To assess CDAI (Clinical Disease Activity Index) score for efficacy
Change from baseline for the HAQ-DI | Baseline to Up to Week 16
  To assess HAQ-DI (Health Assessment Questionnaire - Disability Index) for efficacy
Safety assessed by incidence of adverse events | Up to Week 16
  Adverse events will be coded using Medical Dictionary for Regulatory Activities (MedDRA).
Safety assessed by laboratory tests: Hematology | Up to Week 16
  To assess hematology as a criteria of safety variables.
Safety assessed by laboratory tests: Biochemistry | Up to Week 16
  To assess Biochemistry as a criteria of safety variables.
Safety assessed by laboratory tests: Urinalysis | Up to Week 16
  To assess Urinalysis as a criteria of safety variables.
Safety assessed by vital signs: Body temperature | Up to Week 16
  To assess the vital sign as a criteria of safety variables.
Safety assessed by vital signs: Sitting blood pressure | Up to Week 16
  To assess the vital sign as a criteria of safety variables.
Safety assessed by vital signs: pulse rate | Up to Week 16
  To assess the vital sign as a criteria of safety variables.
Safety assessed by weight | Up to Week 16
  To assess the weight as a criteria of safety variables.
Safety assessed by standard 12-lead electrocardiogram | Up to Week 16
  To assess the cardiovascular system functioning as a criteria of safety variables.
Serum concentration of ASP5094 | Up to Week 16
  To assess Serum concentration of ASP5094 for pharmacokinetics
Serum concentration of TNF-α | Up to Week 16
  To assess TNF-α (Tumor Necrosis Factor-α) for pharmacodynamics
Serum concentration of MMP3 | Up to Week 16
  To assess MMP3 (Matrix metalloproteinase 3) for pharmacodynamics
Serum concentration of IL-6 | Up to Week 16
  To assess IL-6 (Interleukin-6) for pharmacodynamics
Anti-ASP5094 anti-bodies | Up to Week 16
  To assess Anti-ASP5094 anti-bodies for immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (31):
- Japan (31):
  - Site JP00002, Asahikawa
  - Site JP00027, Asahikawa
  - Site JP00029, Beppu
  - Site JP00015, Chiba
  - Site JP00008, Fukuoka
  - Site JP00009, Fukuoka
  - Site JP00026, Fukuoka
  - Site JP00016, Ichinomiya
  - Site JP00012, Kanuma
  - Site JP00028, Kawachi-Nagano
  - Site JP00005, Kitamoto
  - Site JP00025, Kobe
  - Site JP00030, Kobe
  - Site JP00010, Kumamoto
  - Site JP00006, Kyoto
  - Site JP00018, Meguro City
  - Site JP00020, Nagano
  - Site JP00014, Nagoya
  - Site JP00022, Okayama
  - Site JP00011, Ōita
  - Site JP00003, Ōsaki
  - Site JP00019, Sagamihara
  - Site JP00007, Sanuki
  - Site JP00001, Sapporo
  - Site JP00023, Shimonoseki
  - Site JP00021, Shizuoka
  - Site JP00004, Takasaki
  - Site JP00017, Tomakomai
  - Site JP00013, Toyohashi
  - Site JP00024, Tsukuba
  - Site JP00031, Yokohama

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Takeuchi T, Tanaka Y, Erdman J, Kaneko Y, Saito M, Higashitani C, Smulders R, Lademacher C. ASP5094, a humanized monoclonal antibody against integrin alpha-9, did not show efficacy in patients with rheumatoid arthritis refractory to methotrexate: results from a phase 2a, randomized, double-blind, placebo-controlled trial. Arthritis Res Ther. 2020 Oct 21;22(1):252. doi: 10.1186/s13075-020-02336-3. PMID 33087159
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=348